CLINICAL TRIAL: NCT05730608
Title: Improving Breast Cancer Staging With 18F-FDG PET/CT Imaging (The IMBRECAS PET Study)
Brief Title: 18F-FDG PET/CT Imaging for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 495077
Record Dates: First submitted 2023-01-27; First posted 2023-02-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female; Breast Cancer Recurrent

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary breast cancer (Other): Patients diagnosed with new breast cancer determined to have "high risk" disease by a multidisciplinary team.
  Interventions: Other: 18F-FDG PET/CT
- Recurrent breast cancer (Other): Patients with suspected or proven locoregional recurrent breast cancer.
  Interventions: Other: 18F-FDG PET/CT

INTERVENTIONS:
Other: 18F-FDG PET/CT — Included breast cancer patients will undergo a 18F-FDG PET/CT scan in addition to conventional imaging with CT and bone scintigraphy.

SUMMARY:
Purpose To investigate the ability of 18F-FDG PET/CT imaging to detect metastases not detected by conventional imaging (CT and bone scintigraphy) in patients diagnosed with stage II/III and locoregional recurrent breast cancer (BC) which can affect the choice of treatment.

Hypothesis The hypothesis is that 18F-FDG PET/CT can provide information about disease stage beyond the currently used conventional imaging (CT and bone scintigraphy) in patients diagnosed with stage II/III or locoregional recurrent BC.

Objectives

Primary:

To evaluate if a 18F-FDG PET/CT scan in the initial work up of patients diagnosed with stage II/III or locoregional recurrent BC will lead to change in staging and/or treatment.

Secondary:

* Overall survival (OS) and progression-free survival (PFS) in the patients with upstaging based on findings on 18F-FDG PET/CT scan compared with the patients with unchanged stage of disease following 18F-FDG PET/CT.
* Obtain size of the primary BC from CT/MRI scan and evaluate if these metrics are correlated to outcome.
* Obtain PET parameters from the primary BC: maximum, mean, and peak standardized uptake value (SUVmax, SUVmean, SUVpeak), metabolic tumour volume (MTV), total lesion glycolysis (TLG), total MTV and total TLG and evaluate if these metrics are correlated with outcome.
* Obtain CT and PET texture parameters from the primary BC and evaluate if these metrics are correlated with outcome.
* Blood and tumor samples for molecular characterisation:

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk primary or recurrent breast cancer
* Non pregnant women > 18 years
* Not receiving active treatment of other cancer types.
* Eastern Cooperative Oncology Group (ECOG) status 0-2.

Exclusion Criteria:

* Pregnant woman
* Males
* Age under 18
* Patients receiving active treatment for other cancers
* Poor general conditipon (ECOG 3 or higher)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in staging and/or management due to added 18F-FDG PET/CT scan | 5 years
  Percentage of the patients with change in staging and/or management

SECONDARY OUTCOMES:
Overall survival | 5 years
  Survival after 18F-FDG PET/CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Harald Grut, MD, PHD, Principal Investigator — Vestre Viken Hospital Trust
Locations (1):
- Drammen Hospital - Vestre Viken HF, Drammen, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD available by request (Harald Grut, harald.grut@gmail.com)
Supporting Information: Study Protocol, ICF
Time Frame: 10.02.23 to 31.12.32
Access Criteria: IPD available by request (Harald Grut, harald.grut@gmail.com)